CLINICAL TRIAL: NCT03461991
Title: Correlation Between In-vivo Anatomy of Corneal Dystrophies as Assessed by High- Resolution Optical Coherence Tomography (OCT) Measurement and Histological Examination - A Pilot Study
Brief Title: Correlation Between In-vivo Anatomy of Corneal Dystrophies as Assessed by High- Resolution Optical Coherence Tomography (OCT) Measurement and Histological Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPHT-270617
Record Dates: First submitted 2018-01-02; First posted 2018-03-12 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2022-04

CONDITIONS: Corneal Dystrophy
MeSH Terms: conditions — Corneal Dystrophies, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients scheduled for corneal transplantation (Other)
  Interventions: Device: Ultrahigh resolution Spectral Domain OCT

INTERVENTIONS:
Device: Ultrahigh resolution Spectral Domain OCT — A spectrometer based ultrahigh resolution Spectral Domain OCT (SDOCT) system operating at 800 nm for the anterior chamber will be employed in the present study. The spectrum of the Ti:Sapphire laser light source is centered at 800 nm. With a full width at half maximum bandwidth of 170 nm, the axial resolution is 1.3 μm in the cornea. The transverse resolution of the employed OCT system is 21 μm at the front surface of the cornea. For measurement, patients will place their head in a modified slit lamp head rest. During the measurement period, patients will be asked to look straight forward onto an internal fixation target and to avoid blinking. Different scattering patterns, e.g. raster, circular and spiral scans will be employed.

SUMMARY:
Corneal dystrophies are usually classified histopathologically according to the layer of the cornea that is affected. The International Committee for the Classification of Corneal Dystrophies (IC3D) takes this anatomical classification as referral with summarizing clinical, genetic, and pathological data.

Most of this classification relies on slit lamp findings or histologic specimen, since in-vivo imaging of corneal microstructures has only become available in the recent years. With confocal microscopy it is possible to image corneal microstructures at a high resolution, but this technique is limited by its reduced repeatability and the fact that only a small area can be imaged. By the use of optical coherence tomography (OCT) systems it is possible to overcome these limitations. Commercially available systems, however, only have an axial resolution of about 18 µm which is not sufficient for imaging of all corneal layers.

Recently, a high-resolution optical coherence tomography (OCT) system was developed at the Center for Medical Physics and Biomedical Engineering that enables a resolution of about 1 µm. With this resolution, all corneal structures and several pathologies can be visualized.

In the present study the investigators want to use this OCT system to image corneal dystrophies in patients scheduled for corneal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Presence of corneal dystrophy
* Scheduled for corneal transplantation (PK, ALK, DALK, DSAEK or DMEK)
* No previous corneal surgery in the study eye

Exclusion Criteria:

* Participation in a clinical trial in the previous 3 weeks
* Presence of any abnormalities preventing reliable measurements as judged by the investigator
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Correlation in measurement of corneal layers in preoperative high-resolution OCT and histological diagnosis of corneal dystrophies of the removed cornea | preoperative
  Preoperative high-resolution OCT measurement of the corneal layers in the study eye will be performed to assess corneal dystrophies. The corneal tissue removed during surgery will then be sent to the Institute for Clinical Pathology for histological preparation and diagnosis of corneal dystrophies. The correlation between the preoperative measurement and histological diagnosis will be shown to assess the accuracy of measuring corneal layers in high-resolution OCT imaging.

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Vienna
  - Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna

IPD SHARING:
Plan to Share IPD: No